CLINICAL TRIAL: NCT01960439
Title: Responsiveness of Endoscopic Evaluation of Ulcerative Colitis Using a Central Reader Based Image Management System
Brief Title: Responsiveness of Endoscopic Evaluation in UC
Status: Completed | Type: Observational
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: RP1302
Record Dates: First submitted 2013-09-26; First posted 2013-10-10 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Ulcerative Colitis
Keywords: disease activity; central reader; endoscopic indices
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic evaluation: The study population contained a broad spectrum of endoscopic disease and clinical activity. At entry to the trial patients had active disease defined by the presence of a modified UCDAI score between 4 and 10.1 Only patients who had a MMCS endoscopy subscale score according to a single central reader (n= 194 of 281 participants) were eligible for assessment in the current study.

SUMMARY:
The purpose of this study of this study is to assess the responsiveness and validity of CIMS (Central Image Management System)-based endoscopic evaluation of UC (Ulcerative Colitis) clinical disease activity by measuring:

The responsiveness central reader endoscopic EIs [(Endoscopic Indices) (MMCS (Modified Mayo Clinic endoscopy Subscore), UCEIS (Ulcerative Colitis Endoscopic Index of Severity) MBS (Modified Baron Score)] to clinical change from baseline to week 6 in a prospective trial of a treatment of known efficacy in UC.

DETAILED DESCRIPTION:
This study will evaluate the responsiveness central reader based EIs for assessing clinical disease activity. Endoscopic images will be obtained from recent large multicenter randomized clinical trial and assessed using utilizing CIMS readers using EIs (MMCS, UCEIS, MBS) and a VAS (visual analog scale). The primary efficacy endpoint of this trial was clinical and endoscopic remission at week 6, with a secondary endpoint of endoscopic and clinical remission at week 10. For the same subjects, clinical data will be obtained including a modified UCDAI (Ulcerative Colitis Disease Activity Index). Central readers are blinded to clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* Active ulcerative colitis disease defined by the presence of a modified UCDAI score between 4 and 10
* Only patients who had an MMCS endoscopy subscale score according to a single reader
* Endoscopic videos recorded for CIMS based central reader assessment

Exclusion Criteria:

* UCDAI score less than 4 and greater than 10

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population contained a broad spectrum of endoscopic and clinical activity. At entry patients had active disease defined by the presence of a modified UCDAI score between 4 and 10.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Central Reading | 2 years
  Each of 4 central readers will score approximately 130 videos

SECONDARY OUTCOMES:
Endoscopic Responsiveness of endoscopic index to Clinical Change | 2 years
  The effect size of each endoscopic index will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feagan, MD, Principal Investigator — Western University
Locations (1):
- Robarts Clinical Trials Inc., London, Ontario, Canada

REFERENCES:
- [Background] Feagan BG, Sandborn WJ, D'Haens G, Pola S, McDonald JWD, Rutgeerts P, Munkholm P, Mittmann U, King D, Wong CJ, Zou G, Donner A, Shackelton LM, Gilgen D, Nelson S, Vandervoort MK, Fahmy M, Loftus EV Jr, Panaccione R, Travis SP, Van Assche GA, Vermeire S, Levesque BG. The role of centralized reading of endoscopy in a randomized controlled trial of mesalamine for ulcerative colitis. Gastroenterology. 2013 Jul;145(1):149-157.e2. doi: 10.1053/j.gastro.2013.03.025. Epub 2013 Mar 22. PMID 23528626
- [Background] TRUELOVE SC, WITTS LJ. Cortisone in ulcerative colitis; final report on a therapeutic trial. Br Med J. 1955 Oct 29;2(4947):1041-8. doi: 10.1136/bmj.2.4947.1041. No abstract available. PMID 13260656
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095